CLINICAL TRIAL: NCT04542291
Title: Targeting Pancreatic Cancer With Sodium Glucose Transporter 2 (SGLT2) Inhibition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202011019; 1P50CA196510-01A1 (NIH)
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2023-01-17 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Pancreas Cancer; Pancreatic Cancer; Cancer of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Dapagliflozin (Experimental): * Dapagliflozin is an oral drug which will be administered on an outpatient basis. Dosing will start at 5 mg daily and will increase to 10 mg daily after 2 weeks (after consulation with a study endrocrinologist) if the patient is tolerating the 5 mg dose. Dapagliflozin will be given for a total of 8 weeks (2 weeks at 5 mg and 6 weeks at 10 mg)
  * Treatment with dapagliflozin will be initiated on Cycle 1 Day 1 of standard of care chemotherapy.
  * Participants will use the BIOSENSE meter once daily
  Interventions: Drug: Dapagliflozin; Device: BIOSENSE meters

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin will be provided for this trial
  Other Names: Farxiga
Device: BIOSENSE meters — -Being used in this trial to evaluate utility for assessing breath ketones

SUMMARY:
This is a first-in-human, pilot study of the feasibility and safety of dapagliflozin (in addition to standard of care treatment) for the treatment of patients with metastatic pancreatic ductal adenocarcinoma. The primary hypothesis is that dapagliflozin is well-tolerated and safe to use in this patient population. The investigators also hypothesize that dapagliflozin will be efficacious as an adjunct to front-line chemotherapy assessed by decreased tumor markers mediated by its pleiotropic metabolic effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or locally advanced pancreatic ductal adenocarcinoma, pancreatic adenosquamous carcinoma or squamous cell carcinoma
* Patients with treated/stable brain metastases, defined as patients who have received prior therapy for their brain metastases and whose CNS disease is radiographically stable at study entry, are eligible.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* No prior systemic therapy for pancreatic ductal adenocarcinoma in the metastatic or locally advanced setting.
* Planning to receive treatment with nab-paclitaxel and gemcitabine.
* At least 18 years of age.
* ECOG performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Estimated glomerular filtration rate eGFR ≥ 30 mL/min/1.73m^2
* Because chemotherapeutic agents such as nab-paclitaxel and gemcitabine are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and at least one month after completion of the study
* Agreement to adhere to Lifestyle Considerations throughout study duration
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* History of total pancreatectomy
* Current or previous treatment with SGLT2i or thiazolidinedione.
* Currently receiving regularly scheduled systemic steroids in the form of prednisone or dexamethasone. Note that dexamethasone that can be prescribed for nausea on the day of chemotherapy, but in subsequent days will be replaced by a nonsteroidal anti-emetic for patients in this trial. Topical steroid ointments or creams for occasional skin rash is allowed.
* A history of other malignancy with the exceptions of malignancies for which all treatment was completed at least 2 years before registration with no evidence of disease and locally treated skin squamous or basal cell carcinoma.
* History of stroke or transient ischemic attack (in the last 5 years).
* HbA1c > 10% unless approved by endocrinologist
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to dapagliflozin, nab-paclitaxel, gemcitabine or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, peripheral arterial disease, ketoacidosis, severe kidney disease (estimated glomerular filtration rate eGFR < 30 mL/min/1.73m2), symptomatic hypotension, and chronic/frequent urinary tract infections or yeast infections.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kian-Huat Lim, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park LK, Lim KH, Volkman J, Abdiannia M, Johnston H, Nigogosyan Z, Siegel MJ, McGill JB, McKee AM, Salam M, Zhang RM, Ma D, Popuri K, Chow VTY, Beg MF, Hawkins WG, Peterson LR, Ippolito JE. Safety, tolerability, and effectiveness of the sodium-glucose cotransporter 2 inhibitor (SGLT2i) dapagliflozin in combination with standard chemotherapy for patients with advanced, inoperable pancreatic adenocarcinoma: a phase 1b observational study. Cancer Metab. 2023 May 18;11(1):6. doi: 10.1186/s40170-023-00306-2. PMID 37202813
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin
Started | 15
Completed | 12
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 68 [57 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Tolerability as Measured by Number of Participants With Related Adverse Events
Description: * Adverse events will be graded with CTCAE v. 5.0.
  * Related indicates adverse events possibly, probably, or definitely related to treatment.
Time Frame: From start of treatment through 30 days after treatment (estimated to be 3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 15
Participants
  Anemia | 15
  Atrial fibrillation | 1
  Colitis | 1
  Constipation | 1
  Diarrhea | 6
  Dry mouth | 1
  Nausea | 5
  Vomiting | 3
  Chills | 2
  Edema limbs | 2
  Fatigue | 6
  Fever | 2
  Sepsis | 1
  Skin infection | 1
  Alanine aminotransferase increased | 8
  Alkaline phosphatase increased | 5
  Aspartate aminotransferase increased | 6
  Lymphocyte count decreased | 7
  Neutrophil count decreased | 7
  Platelet count decreased | 12
  White blood cell decreased | 10
  Anorexia | 5
  Hypoalbuminemia | 2
  Hyponatremia | 2
  Dysgeusia | 1
  Headache | 1
  Peripheral sensory neuropathy | 4
  Chronic kidney disease | 2
  Proteinuria | 1
  Alopecia | 11
  Hyperhidrosis | 1
  Pruritus | 1
  Rash maculo-papular | 2
  Rash on arm | 1
  Hypotension | 1

2. Secondary Outcome: Changes in Plasma Glucose
Time Frame: Screening, Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, and End of Treatment (estimated to be 2 months)
Population: The three patients who did not complete treatment are not evaluable for this outcome measure.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 12
mg/dL
  Screening | 110 [71 to 158]
  Cycle 1 Day 1 | 106.5 [74 to 138]
  Cycle 1 Day 15 | 108.5 [79 to 138]
  Cycle 2 Day 1 | 100.5 [79 to 164]
  Cycle 2 Day 15 | 102.5 [82 to 172]
  End of Treatment | 98 [81 to 195]

3. Secondary Outcome: Changes in Ketones
Description: -Patients are to collect and test ketones weekly while on treatment.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 22, Cycle 2 Day 1, Cycle 2 Day 8, Cycle 2 Day 15, and Cycle 2 Day 22
Population: The three patients who did not complete treatment are not included in this outcome measure and an additional patient is not included as they didn't collect any ketone readings. There are additional patients who missed ketone readings at additional time points.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 11
mg/dL
  Cycle 1 Day 1: number analyzed (Participants) | 10
  Cycle 1 Day 1 | 0.5 [0 to 5]
  Cycle 1 Day 8: number analyzed (Participants) | 9
  Cycle 1 Day 8 | 0 [0 to 5]
  Cycle 1 Day 15 | 0 [0 to 5]
  Cycle 1 Day 22 | 0 [0 to 5]
  Cycle 2 Day 1: number analyzed (Participants) | 10
  Cycle 2 Day 1 | 0 [0 to 5]
  Cycle 2 Day 8: number analyzed (Participants) | 9
  Cycle 2 Day 8 | 0 [0 to 5]
  Cycle 2 Day 15: number analyzed (Participants) | 9
  Cycle 2 Day 15 | 0 [0 to 5]
  Cycle 2 Day 22: number analyzed (Participants) | 7
  Cycle 2 Day 22 | 0 [0 to 5]

4. Secondary Outcome: Changes in HbA1c
Time Frame: Screening and Cycle 2 Day 15
Population: The three patients who did not complete treatment are not evaluable for this outcome measure.
Measure: Median (Full Range); unit: percentage of glycosylated hemoglobin
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 12
percentage of glycosylated hemoglobin
  Screening | 5.95 [4.2 to 7.2]
  Cycle 2 Day 15 | 5.95 [5.2 to 7.2]

5. Secondary Outcome: Changes in CA19-9
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, and End of Treatment, up to 8 weeks
Population: The three patients who did not complete treatment are not evaluable for this outcome measure. There are 3 additional patients not evaluable for this outcome measure because 2 patients did not have detectable levels of CA19-9 prior to treatment and 1 patient did not have the end of treatment CA19-9 drawn.
Measure: Median (Full Range); unit: U/mL
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 9
U/mL
  Cycle 1 Day 1 | 1060 [27.3 to 25010]
  Cycle 2 Day 1 | 315.6 [23.3 to 9250]
  End of Treatment | 256.1 [11.3 to 30330]

6. Secondary Outcome: Changes in Total Fat Volume in Visceral Fat Area as Assessed by CT-based Body Composition
Time Frame: From pre-treatment and post-8 weeks of treatment
Population: The three patients who did not complete treatment are not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 12
cm^3
  Pre-treatment | 5009.845557 (1894.271988)
  Post-8 weeks of treatment | 4334.134004 (2127.102525)

7. Secondary Outcome: Changes in Total Skeletal Muscle Volume in Visceral Fat Area as Assessed by CT-based Body Composition
Time Frame: From pre-treatment and post-8 weeks of treatment
Population: The three patients who did not complete treatment are not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 12
cm^3
  Pre-treatment | 1494.813884 (324.0522377)
  Post-8 weeks of treatment | 1360.211117 (315.4997407)

8. Secondary Outcome: Changes in Total Muscle to Fat Ratio in Visceral Fat Area as Assessed by CT-based Body Composition
Time Frame: From pre-treatment and post-8 weeks of treatment
Population: The three patients who did not complete treatment are not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 12
ratio
  Pre-treatment | 0.378776105 (0.274872687)
  Post-8 weeks of treatment | 0.518539627 (0.638171644)

9. Secondary Outcome: Changes in CT-quantified Tumor Size
Time Frame: From pre-treatment and post-8 weeks of treatment
Population: The three patients who did not complete treatment are not evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 12
cm
  Pre-treatment | 7.541666667 (4.825775177)
  Post-8 weeks of treatment | 7.358333333 (5.946038916)

10. Secondary Outcome: Change in Tumor Necrosis
Time Frame: From pre-therapy to post-8 weeks of therapy
Population: The CT scans were unable to determine the scope of tumor necrosis.
Arm/Group | Dapagliflozin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days after discontinuation of dapagliflozin. Treatment was 8 weeks in length. All-cause mortality was collected from start of treatment through completion of follow-up. Follow-up was an additional 3 months after completion of treatment.
Arm/Group | Dapagliflozin
All-Cause Mortality (participants affected / at risk) | 10/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=15)
Atrial fibrillation (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Sepsis (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=15)
Anemia (Blood and lymphatic system disorders) | 15
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Rectal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 7
Disease progression (General disorders) | 3
Edema limbs (General disorders) | 7
Fatigue (General disorders) | 6
Fever (General disorders) | 3
Biliary tract infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Salmonella enteritis infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Burn (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 7
Anorexia (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 6
Blood bicarbonate increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 12
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 10
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 7
Arthalgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Calf pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 3
Glucosuria (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 11
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Nail changes (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Peeling of feet (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Rash on arm (Skin and subcutaneous tissue disorders) | 1
Redness in left leg (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04542291/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04542291/ICF_000.pdf